CLINICAL TRIAL: NCT00005647
Title: A Phase I Pharmacokinetic, Pharmacodynamic, and Clinical Study of the Combination of the Angiogenesis Inhibitor SU5416 and Paclitaxel in Recurrent or Metastatic Carcinoma of the Head and Neck
Brief Title: SU5416 and Paclitaxel in Treating Patients With Recurrent, Locally Advanced or Metastatic Cancer of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1399; U01CA062502 (NIH); P30CA043703 (NIH); CWRU-1399; NCI-T99-0084
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Head and Neck Cancer
Keywords: thyroid gland medullary carcinoma; anaplastic thyroid cancer; recurrent thyroid cancer; recurrent salivary gland cancer; recurrent metastatic squamous neck cancer with occult primary; stage III follicular thyroid cancer; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent hypopharyngeal cancer; stage III adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Medullary; Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms; Salivary Gland Neoplasms; Adenocarcinoma, Follicular; Hypopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory | interventions — Paclitaxel; Semaxinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: paclitaxel — Patients receive paclitaxel IV over one hour on day 1. Treatment continues weekly in the absence of disease progression or unacceptable toxicity.
Drug: semaxanib — Patients receive SU5416 IV over one hour on days 1 and 4. Treatment continues weekly in the absence of disease progression or unacceptable toxicity.
  Other Names: SU5416

SUMMARY:
RATIONALE: SU5416 may stop the growth of head and neck cancer by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining SU5416 with chemotherapy may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of SU5416 and paclitaxel in treating patients who have recurrent, locally advanced, or metastatic cancer of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and safety of SU5416 and paclitaxel in patients with recurrent or metastatic head and neck cancer.
* Determine the antiangiogenesis effect of this combination regimen in these patients.
* Determine the toxicity, pharmacodynamic effects, and pharmacokinetic parameters of this combination.

OUTLINE: This is a dose escalation study.

Patients receive paclitaxel IV over one hour on day 1 and SU5416 IV over one hour on days 1 and 4. Treatment continues weekly in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paclitaxel and SU5416 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose limiting toxicities.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study within 9-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Metastatic or loco-regionally recurrent malignancy of the head and neck (including salivary gland and thyroid) that is incurable by surgery or radiotherapy
* At least two distinct tumor masses OR
* One tumor mass at least 3 cm in diameter
* No brain metastases
* No pulmonary metastases as only site of disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm3
* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin greater than 9.0 g/dL

Hepatic:

* PT and PTT normal OR
* INR ratio less than 1.1
* Bilirubin less than 1.5 mg/dL
* AST and ALT less than 2 times upper limit of normal

Renal:

* Creatinine less than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No uncompensated coronary artery disease
* No history of myocardial infarction or severe or unstable angina within the past 6 months
* No severe peripheral vascular disease
* No deep venous thrombosis or arterial thrombosis within the past 6 months
* No known hypercoagulable syndrome with predisposition to venous or arterial clots

Pulmonary:

* No pulmonary embolism within the past 6 months

Other:

* No prior cerebral hemorrhage
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since palliative chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* At least 4 weeks since combined chemoradiotherapy and recovered
* Must be recovered from prior taxanes

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior large field radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-05; Primary Completion 2002-12 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and safety of SU5416 and paclitaxel. | Treatment continues weekly in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States